CLINICAL TRIAL: NCT01094587
Title: Sutureless vs Sutured Gastroschisis Closure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulty
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matias Bruzoni, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-10142009-4180; IRB Protocol: 16918
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Gastroschisis
MeSH Terms: conditions — Gastroschisis | interventions — Sutures

ARMS (2):
- Sutured closure (Active Comparator)
  Interventions: Procedure: Gastroschisis closure with suture
- Sutureless closure (Active Comparator)
  Interventions: Procedure: Gastroschisis closure without suture

INTERVENTIONS:
Procedure: Gastroschisis closure with suture
  Arms: Sutured closure
Procedure: Gastroschisis closure without suture
  Arms: Sutureless closure

SUMMARY:
This study aims to prospectively assess outcomes of sutureless versus sutured gastroschisis closure with a randomized control trial. The parameters of this trial were determined using our retrospective study as pilot data. Primary outcome measures will be time on ventilator and time to initiating enteral feeds. Other outcome measures will include cosmetic outcome, length of hospital stay and the associated rate of complications, including bowel resection, sepsis, and death.

DETAILED DESCRIPTION:
This study aims to prospectively assess outcomes of sutureless versus sutured gastroschisis closure with a randomized control trial. The parameters of this trial were determined using our retrospective study as pilot data. Primary outcome measures will be time on ventilator and time to initiating enteral feeds. Other outcome measures will include cosmetic outcome, length of hospital stay and the associated rate of complications, including bowel resection, sepsis, and death.

In comparing these techniques of gastroschisis closure, we can further evaluate which is the safer and more efficacious method, thereby improving patient care while decreasing hospital cost.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria are the diagnosis of gastroschisis, birth weight of 1500 grams or greater, and gestational age of 34 weeks or more.

Exclusion Criteria:Exclusion criteria are infants with other major abnormalities or medical conditions, grade IV intraventricular hemorrhage, inability to obtain informed consent, and the presence of a closed-type gastroschisis defect.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2015-06-24 (Actual); Study Completion 2015-06-24 (Actual)

PRIMARY OUTCOMES:
Time on ventilator | Up to 1 week
Time to initiating enteral feeds | Up to 4 weeks

SECONDARY OUTCOMES:
Cosmesis | 6 months after hospital discharge
Length of hospital stay | Up to 6 weeks
Complications including bowel resection, sepsis, and death. | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Dutta, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States